CLINICAL TRIAL: NCT06843005
Title: Serial Coronary CTA-based Plaque Progression Detection for Management of Coronary Heart Disease: a Randomised Controlled Trial
Brief Title: Serial Coronary CTA-based Plaque Progression Detection for Management of Coronary Heart Disease
Acronym: SUCCESS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zhang longjiang,MD (Other)
Responsible Party: Sponsor-Investigator, Zhang longjiang,MD, Principal Investigator : Zhang longjiang, Jinling Hospital, China
Organization: Jinling Hospital, China (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2024DZKY-132-01
Record Dates: First submitted 2025-02-14; First posted 2025-02-24 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-03

CONDITIONS: Major Adverse Cardiovascular Events (MACE); Prevention; Coronary Artery Disease(CAD); CT Angiography
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CCTA-based follow-up management group (Active Comparator): The subjects will undergo routine clinical and laboratory examinations, as well as follow-up CCTA examinations to assess the progression of plaques and to recommend appropriate management, treatment, and follow-up based on the findings
  Interventions: Diagnostic Test: Coronary Computed Tomography Angiography
- clinical-based follow-up management group (Sham Comparator): The subjects will undergo routine clinical and laboratory examinations, and recommendations for appropriate management, treatment, and follow-up will be made based on the results.
  Interventions: Other: Current clinical guidelines

INTERVENTIONS:
Diagnostic Test: Coronary Computed Tomography Angiography — Based on the assessment of plaque progression after follow-up CCTA examination, patients will be given either intensive treatment or routine treatment.
  Arms: CCTA-based follow-up management group
Other: Current clinical guidelines — Patients will be treated according to the 2024 ESC Guidelines for the Management of Chronic Coronary Syndromes.
  Arms: clinical-based follow-up management group

SUMMARY:
The primary objective of this study is to evaluate whether a management strategy based on coronary computed tomography angiography (CCTA) for patients with non-obstructive coronary artery disease can improve the LDL-C target achievement rate compared to a traditional management strategy without follow-up CCTA, thereby reducing the incidence of major adverse cardiovascular and cerebrovascular events over a 3 years period, including all-cause mortality, myocardial infarction, ischemia driven revascularation and stroke.

DETAILED DESCRIPTION:
Patients with non-obstructive coronary artery disease have a high rate of adverse cardiovascular events, and currently, there is still a lack of effective management strategies for these patients in clinical practice. In the SUCCESS study, investigator will compare follow-up CCTA management with routine clinical management to assess the effectiveness of follow-up CCTA in improving lipid control and reducing cardiovascular events in these patients.

The SUCCESS study is a single-center, randomized, parallel-controlled, interventional clinical trial that recruits patients with non-obstructive coronary artery disease identified on previous CCTA (coronary artery stenosis of 20% to 70% or left main coronary artery stenosis of 20% to 50%). The experimental group is the CCTA follow-up management group, and the control group is the routine clinical follow-up management group. All participants will be randomly assigned to the experimental and control groups in a 1:1 ratio. The experimental group will undergo management using follow-up CCTA, while the control group will be managed using routine clinical and laboratory examinations. At the 1-year follow-up, all participants will undergo laboratory re-examination to observe the impact of follow-up CCTA on lipid target achievement. After 3 years of follow-up, the differences in the occurrence of major adverse cardiovascular and cerebrovascular events (MACCE) between the two groups will be compared.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 80 years old;
2. Known patients with non-obstructive coronary artery disease (disease duration ≥2 years);
3. Patients who agree to undergo follow-up CCTA examinations and cooperate in completing follow-up observations.

Exclusion Criteria:

1. Patients who have experienced ACS or PCI/CABG;
2. Patients who have experienced adverse cardiovascular and cerebrovascular events;
3. Patients who have undergone follow-up CCTA or DSA examinations before enrollment;
4. Patients with severe hepatic and renal dysfunction;
5. Patients with contraindications to CCTA examinations;
6. Patients with poor initial CCTA image quality or data loss.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3100 (Estimated)
Dates: Start 2025-02-28 (Actual); Primary Completion 2028-12-30 (Estimated); Study Completion 2028-12-30 (Estimated)

PRIMARY OUTCOMES:
Major adverse cardiovascular and cerebrovascular event | 36 months after baseline
  Record the number of participants experiencing major adverse cardiovascular and cerebrovascular event such as all-cause mortality, non-fatal myocardial infarction, ischemia driven revascularation and stroke

SECONDARY OUTCOMES:
LDL-C control rate | 12 months after baseline
  The proportion of participants with controlled LDL-C（<1.4mmol/L）
Mean LDL-C changes | 12 months after baseline
  Mean LDL-C changes of participants
Adherence to lipid-lowering medication rate | 12 months after baseline
  The proportion of participants who adhere to lipid-lowering drugs
The difference in healthcare-seeking rates between the two groups | 12 months after baseline
  The difference in healthcare-seeking rates between the two groups of patients, including both regular follow-ups and visits driven by clinical symptoms of coronary heart disease
Hypertension control rate | 12 months after baseline
  The proportion of participants with SBP<140mmHg and DBP<90mmHg.
Diabetic control rate | 12 months after baseline
  The proportion of participants with HbA1c <53 mmol/mol (7.0%).
Cardiac death | 36 months after baseline
  Number of participants diagnosed with cardiovascular death
Fatal and non-fatal myocardial infarction or stroke | 36 months after baseline
  Number of participants diagnosed with myocardial infarction or stroke
Rehospitalization due to progressive angina | 36 months after baseline
  Number of patients seeking medical care for unstable angina
Major adverse cardiovascular event | 36 months after baseline
  Record the number of participants experiencing major adverse cardiovascular events such as all-cause mortality, non-fatal myocardial infarction and ischemia driven revascularation
Procedures | 36 months after baseline
  The proportion of participants undergone procedures，including Invasive coronary angiography, percutaneous coronary intervention and coronary artery bypass graft surgery
Radiation dose and incidental findings from CTCA | 36 months after baseline
  The total radiation dose received by the participants during multiple examinations after enrollment.
Change in quality of life (SF-12) | 36 months after baseline
  Change in quality of life measured using 12-item Short-Form Health Survey Questionnaire (SF-12) instrument
The primary outcome in different subgroups | 36 months after baseline
  The primary outcome (all-cause mortality, non-fatal myocardial infarction, ischemia driven revascularation and stroke) will be analyzed in prespecified subgroups, including age, sex, hypertension, diabetes mellitus, degree of stenosis on baseline CCTA.

CONTACTS AND LOCATIONS:
Overall Officials: Trail Manager, Study Chair — Jinling Hospital,Nanjing University School of Medicine,Nanjing,China
Locations (1):
- Research Institute Of Medical Imaging Jinling Hospital, Nanjing, Jiangsu, China